CLINICAL TRIAL: NCT02626221
Title: A Prospective Non-interventional Study to Collect Real Life Clinical Data on the Impact of Therapy, the Diagnosis and Management of Chronic Urticaria in Patients Refractory to at Least One Course of H1 Antihistamine Therapy
Brief Title: A Worldwide Antihistamine-Refractory Chronic Urticaria Patient Evaluation in Latin America and Canada (AWARE-LACan)
Acronym: AWARE-LACan
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CIGE025EVE01
Record Dates: First submitted 2015-01-15; First posted 2015-12-10 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Chronic Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single: Single Cohort Study
  Interventions: Other: Non Interventional Study

INTERVENTIONS:
Other: Non Interventional Study — Non Interventional Study

SUMMARY:
This is a non-interventional, multi-country, Latin American study utilizing a prospective single-cohort design. Eligible CU patients will be enrolled in the study and will be followed for 24 months (± 6 weeks).

In accordance with the observational nature of the study, there will be no interventions or interference with the routine care of the patient which will be based solely on the clinical judgment of the treating physician. However, with respect to the frequency and schedule of assessments, the schedule included in Table 7-1 will be recommended.

The selection of the treatment for CU will be clearly separated from the decision to include the patient in the study, and will be made at the discretion of the treating physician in accordance with standard medical practice, the investigator's clinical judgment, and global urticarial guidelines.

In order to prevent selection bias, investigators should offer enrollment to all consecutive patients meeting study criteria, likely to be available for the full duration of the follow-up period of 24 months, and willing to participate in the study.

The overall objective of the study is to evaluate in real-life the CU disease burden, the current treatment patterns and the use of health care resources in patients refractory to H1-antihistamine treatment

ELIGIBILITY:
Inclusion Criteria:

Men or Women at least 18 years of age or older. Patient has medically confirmed diagnosis of chronic urticaria present for more than 2 months.

Patient has been treated with at least one course of H1 antihistamines and is refractory to this treatment Patient has provided written informed consent allowing the use of their anonymous data for the purposes of the study

Exclusion Criteria:

Patient is currently participating in a clinical trial. Patient is, in the opinion of the treating physician, unlikely to be available for the full duration of the follow-up period of 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible Latin American Chronic Urticaria adult patients, males and females, with at least one course of H1 antihistamines and is shown to be refractory to this treatment
Sampling Method: Non-Probability Sample
Enrollment: 497 (Actual)
Dates: Start 2014-12-24 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Change in CU-Quality of Life Questionnaire Score | Last 15 days before each visit
  The CU-QoL is a validated instrument with established psychometric properties developed specifically for the assessment of the health burden of CU. The 2013 international CU guideline recommends the use of CU-Q2oL for assessing quality of life impairment and monitoring disease activity.

SECONDARY OUTCOMES:
Angioedema Quality of Life Questionnaire (AE-QoL) | Last 4 weeks before each visit
  For patients with angioedema, the symptom-specific quality of life will be assessed over the course of the study with the Angioedema Quality of Life Questionnaire (AE-QoL)
Change in Dermatology Life Quality Index (DLQI). | Last 7 days before each visit
  A 10-item dermatology-specific health-related quality-of-life measure assessing dermatology symptoms and their impact on various aspects of life, during the course of the study
Urticaria Activity Score for 7 days (UAS7) | Last 7 days before each visit
  Patients willing and able to comply with the UAS7 assessment will be given a paper-based urticaria diary at every site visit and be asked to complete it daily over the week preceding the next site visit. The diary consists of questions to evaluate the severity of their disease, and patients have to assess the severity of their disease, numbers of wheals and severity of itching
Angioedema Activity Score (AAS) | Last 24 hours before each visit
  The Angioedema Activitiy Score (AAS) is a validated, easy to use tool to determine disease activity in patients with recurrent angioedema, independent of its underlying causes. The AAS is designed to be used by patients for their daily documentation of swelling episodes including their duration, severity and impact on daily functioning and appearance.
Urticaria Control Test (UCT) | Last 4 weeks before each visit
  Short questionnaire assessing how well the urticaria symptoms were controlled over the last 4 weeks
6-item Work Productivity and Activity Impairment (WPAI) instrument | Last 7 days before each visit
  Respondents are asked questions about work and activity impairment due to health problems

OTHER OUTCOMES:
Patient demographics | At the baseline
  Information like: (age, gender) and physical characteristics (height, weight).
CU history including the method of diagnosis | At the baseline
  Including diagnostic aids/tools used, ASST results), the time of onset of CU, the CU type (spontaneous, inducible or both), and the prevalence of inducible types of urticaria (e.g. cold, heat, light, aquagenic, cholinergic, contact), if applicable.
The presence of angioedema at baseline and during the course of the study (incidence and number of events). | Every 3 months, for 24 months
  Angioedema is typically characterized by: 1.-Sudden, pronounced swelling of the lower dermis and subcutis. 2.-Sometimes pain rather than itching. 3.-Frequent involvement below mucous membranes. 4.-Up to 72 hours for resolution
Previous and concomitant CU treatments including treatment adjustments during the course of the study. | Every 3 months, for 24 months
  Concomitant medications
Patient-reported use of CU-related health care resources | Every 3 months, for 24 months
  Including hospitalizations (frequency and duration), emergency room visits (frequency), planned and unplanned visits to a physician (frequency), and phone calls.
Incidence of spontaneous disease remission and the time to spontaneous remission | Every 3 months, for 24 months
  As per physician judgment
Proportion of patients responding to each class of therapy | Every 3 months, for 24 months
  As per physician judgment
Changes in the type of CU (spontaneous, inducible, or both) and the types of inducible urticaria | Every 3 months, for 24 months
  As per physician judgment
Patient satisfaction with treatment as assessed on a simple 0-10 VAS scale | Every 3 months, for 24 months
  simple VAS scale where '0' corresponds to poorly satisfy and '10' corresponds to highly satisfy

CONTACTS AND LOCATIONS:
Locations (28):
- Argentina (8):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Lobos, Buenos Aires
  - Novartis Investigative Site, Buenos Aires, Nueve De Julio
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Salta
- Brazil (5):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Alphaville / Barueri, São Paulo
  - Novartis Investigative Site, Guarulhos, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Colombia (4):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bogotá, Cundinamarca
  - Novartis Investigative Site, Medellín
- Costa Rica (2):
  - Novartis Investigative Site, San José
  - Novartis Investigative Site, San Rafael Escazu
- Dominican Republic (3):
  - Novartis Investigative Site, Santiago de los Caballeros, Republica Dominicana
  - Novartis Investigative Site, Santo Domingo, Republica Dominicana
  - Novartis Investigative Site, Santo Domingo
- Novartis Investigative Site, Guatemala City, Guatemala
- Honduras (2):
  - Novartis Investigative Site, San Pedro Sula
  - Novartis Investigative Site, Tegucigalpa
- Novartis Investigative Site, Panama City, Panama
- Peru (2):
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, San Martín de Porres, Lima region

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com